CLINICAL TRIAL: NCT00464295
Title: Phase II Trial of Capecitabine for the Treatment of Unresectable/ Metastatic or Advanced Hepatocellular Carcinoma(HCC)
Acronym: HCC-CAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Muhammad Kashif Anis, Aga Khan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 449-Med/ERC-05
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; Phase 2 Trial; Capecitabine; Treatment Efficacy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capecitabine in HCC

SUMMARY:
In patients with unresectable/advanced Hepatocellular Carcinoma receiving Capecitabin, we anticipate that the proposed chemotherapy will have a delay in progression of the disease . It is also expected that proposed chemotherapy will have acceptable toxicity and Quality of life.

DETAILED DESCRIPTION:
II. OBJECTIVES

II.A. Primary Objectives: To evaluate response rate (RR) and overall survival (OS).

II.B. Secondary Objective: To evaluate the time to progression (TTP), median time to response (MTR), toxicity and quality of life (QOL).

III. STUDY DESIGN:

III.A. Inclusion criteria:

1. Written informed consent. 2. Age between 18 and 70 years. 3. Documented by at least 2 out of three mentioned criteria and evidence of non-resectability.

1. Radiological either CT Scan/US abdomen
2. Biopsy,
3. Serum alphafeto protein level 4. Multi centric hepatoma or TNM Classification Stage IV. 5. Child's class B or C with a Child's score of maximum 11. 6. No other active malignancy except localized basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

   7. Life expectancy of greater then 3 months. 8. Current laboratory values must be within the limits listed below: Haemoglobin > 8 g/dL WBC > 4,000/uL Absolute Neutrophil Count > 1,500/uL Platelets > 75,000/uL 9. ECOG Performance status of < 2. 10. Patients who have received adjuvant or neoadjuvant therapy are eligible. A minimum interval of 4 weeks since last chemotherapy will be required.

   11. Prior radiotherapy will be allowed if it did not involve a site used to assess response and 4 weeks have elapsed since completion of radiotherapy.

   III.B. Exclusion criteria:

   1. History of allergic reaction to compound chemically related to CAP. 2. Concomitant or previous malignancies within five years other than basal or squamous cell carcinoma of the skin and carcinoma in situ of the cervix. 3. Active, uncontrolled infection. . 5. Concurrent medical problems which could limit the life expectancy or the ability of the patient to receive chemotherapy.

   6. Mental condition that could limit the patient in comprehending the concept of clinical trial or complying with its requirements.

   7. Brain or leptomeningeal involvement. 8. Pre-existing neurotoxicity of >=grade 2. 9. Concomitant radiotherapy, unless localised for bone pain control or palliation.

   10. Being of reproductive potential and not agreeing to practice an effective contraceptive method.

   11. Pregnancy or lactation. 12. Severe renal impairment with Creatinine clearance <30ml/minute. 13. Documented Cardiomyopathy or severe coronary artery disease, or history of arrhythmias.

   IV. PATIENT REGISTRATION

   All patients entering this study must be registered by contacting:

   Drs. Kashif Anis/Zaigham Abbas -Research Co-ordinators The Aga Khan University Hospital, Dept of Medicine/ Medical Oncology. Stadium Road, P.O. Box: 3500, Karachi, 74800, Pakistan Tel (021) 493-0051

   V. THERAPY

   This is a Phase II trial studying chemotherapy with CAP in non-resectable HCC. Prior chemotherapy, radiation therapy, surgery is permitted. Staging is required with a CAT scan/Ultrasound of abdomen and bone scan if necessary. Pre study evaluation should include CBC, renal functions assessment, and liver function tests. Patients will require independent evaluation with medical oncologist/gastroenterologist prior to being included in the study. Chemotherapy would be given in cycles of 21 days. CAP would be given as oral tablets twice daily starting from day 1 to day 14. Medication with standard anti-emetics, which may include serotonin antagonist, may be used before administration of chemotherapy. Duration of chemotherapy administration would be determined by the patient's response. A patient who has progressive disease, is not able to tolerate chemotherapy and has unacceptable toxicity would be taken off the study. Patients, who have a response, will continue on chemotherapy till progression of disease or inability to tolerate chemotherapy is documented.

   VI. DOSE MODIFICATION

   Hematologic Toxicity:

   Chemotherapy will be held if ANC < 1,500/uL, and/or platelet count is < 50,000/uL. Treatment will resume when counts recover. Growth factors can be used in subsequent cycles if delay is secondary to neutropenia. If there is no recovery after 3 weeks of delay, the patient will be taken off the study.

   Renal dysfunction:

   Creatinine Clearance mL/min Dose >50 100% 30-50 75% <30 0%(no treatment is given)

   Elevated Liver Function Tests:

   In the event that bilirubin is elevated during the study, the next cycle will be delayed by a maximum of 2 weeks. (The following dose modification in the dose of capecitabine will be made if the AST and/or ALT and/or alkaline phosphatase levels are elevated:

   AST/ALT Alkaline Phosphatase Recommended dose (%) > 1.5- < 2.5 x normal < 2.5 x normal 75% > 2.5- < 5 x normal > 2.5- < 5 x normal 50% > 5 x normal > 5 x normal Dose delay by a maximum of 2 weeks. If no recovery is noted; the patient should go off study.

   Cardio toxicity:

   Significant drop in left ventricular ejection fraction and/or clinical signs and symptoms of cardiac failure will result in discontinuation from the study.

   Dose Modification:

   Dose reduction is planned if significant (Grade III/IV) hematologic or non-hematologic toxicities are observed. CAP shall be reduced by 25% with grade III/IV toxicity occur. Patient should be taken off study if a life threatening complication occurs. All grade III/IV toxicities should be recorded in detail including the dates of onset and resolution/outcome. GI toxicity of grade II including severe diarrhea, nausea, vomiting and stomatitis, dose modification will be done as, it will be held for 1 week along with symptomatic treatment , if no improvement for 2 weeks then patient will be taken off the study.

   VII. SERIOUS ADVERSE EVENT REPORTING

   All serious events (as defined in Appendix E of protocol) must be reported, as soon as you are aware of them to:

   Drs. Kashif Anis/Zaigham Abbas , at the Aga Khan University Hospital VIII. EVALUATION

   Evaluation before Treatment:

   Patient should have evaluation by gastroenterology/oncology to determine eligibility.

   All Patients should have:

   Diagnosis of hepatoma with the help of Biopsy if possible, or by the help of CT Scan or Serum alpha fetoprotein level, fulfilling 2 out of 3 criteria.

   Complete history and physical examination. CBC, differential, platelet count, serum sodium, potassium, glucose, calcium, creatinine, bilirubin, alkaline phosphatase, AST, ALT ,alpha fetoprotein(AFP), prothrombin time PT and Serum Albumin.

   CT scan of the abdomen with contrast. Cardiac evaluation of LVEF CT scans and plain x-rays if clinically indicated.

   Evaluation during Chemotherapy:

   CBC, differential, platelets count, sodium, potassium, creatinine, glucose, bilirubin, alkaline phosphatase, AST/ALT.

   CBC should be repeated prior to every chemotherapy course.

   Re-evaluation of response after every 3 courses of chemotherapy would be done radio logically by repeating a CT scan/x rays as indicated by sites of disease involvement.

   Evaluation After chemotherapy:

   All patients will be followed thereafter cessation of chemotherapy due to progression of disease, every three to six months until a total of five years for evaluation of five-year disease free and overall survival.

   Evaluation of toxicity profile.

   This should be based either on the NCIC common toxicity criteria (attached at the end), or any other major toxicity criteria (e.g. NCI), and documented in the attached form.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age between 18 and 70 years.
* Documented by at least 2 out of three mentioned criteria and evidence of non-resectability.

  1. Radiological either CT Scan/US abdomen
  2. Biopsy,
  3. Serum alphafeto protein level
* Multi centric hepatoma or TNM Classification Stage IV.
* Child's class B or C with a Child's score of maximum 11.
* No other active malignancy except localized basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Life expectancy of greater then 3 months.
* Current laboratory values must be within the limits listed below:

Haemoglobin > 8 g/dL WBC > 4,000/uL Absolute Neutrophil Count > 1,500/uL Platelets > 75,000/uL

* ECOG Performance status of < 2.
* Patients who have received adjuvant or neoadjuvant therapy are eligible. A minimum interval of 4 weeks since last chemotherapy will be required.
* Prior radiotherapy will be allowed if it did not involve a site used to assess response and 4 weeks have elapsed since completion of radiotherapy.

Exclusion Criteria:

* History of allergic reaction to compound chemically related to CAP.
* Concomitant or previous malignancies within five years other than basal or squamous cell carcinoma of the skin and carcinoma in situ of the cervix.
* Active, uncontrolled infection. .
* Concurrent medical problems which could limit the life expectancy or the ability of the patient to receive chemotherapy.
* Mental condition that could limit the patient in comprehending the concept of clinical trial or complying with its requirements.
* Brain or leptomeningeal involvement.
* Pre-existing neurotoxicity of >=grade 2.
* Concomitant radiotherapy, unless localised for bone pain control or palliation.
* Being of reproductive potential and not agreeing to practice an effective contraceptive method.
* Pregnancy or lactation.
* Severe renal impairment with Creatinine clearance <30ml/minute.
* Documented Cardiomyopathy or severe coronary artery disease, or history of arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To evaluate response rate and overall survival after completing minimum of three cycles of Capecitabine in Advance HCC | 12 months from the start of chemotherapy

SECONDARY OUTCOMES:
To evaluate the time to progression, toxicity and quality of life for patients on chemotherapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad K Anis, MD, Principal Investigator — Aga Khan University; Zaigham Abbas, MD, Principal Investigator — Aga Khan University; Wasim Jafri, MD, Study Director — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan